CLINICAL TRIAL: NCT06865573
Title: Reintegration, Coping, and Care of Families After Inpatient Child and Adolescent Psychiatric Treatment
Brief Title: Youth Mental Health Recovery in the Family After Inpatient Stay
Acronym: ReCoVer
Status: Not yet recruiting | Type: Observational
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Amos-Silvio Erik Friedrich, Principal Investigator, University of Vienna
Other Study IDs: 01291
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Burden; Family Characteristics; Parent-Child Interactions
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- caregivers: primary caregivers of youth who received inpatient psychiatric treatment

SUMMARY:
The goal of this longitudinal mixed-methods study is to investigate caregiver strain, family processes and health outcomes after youth psychiatric inpatient treatment. Caregivers of youth who received inpatient treatment for mental health problems will complete a survey at three timepoints (baseline, 3- and 6- month followup) reporting on youth outcomes, caregiver well-being, and family processes. Qualitative interviews on caregivers' challenges, needs, and resources around the return to home care are conducted with a subsample (target n = 10) of participants.

The main research questions (RQs) are:

RQ 1: Do family processes contribute to youth mental health outcomes after discharge from inpatient treatment? RQ 1a: What family-level risk factors predict youth readmission to inpatient treatment? RQ 1b: Do family processes predict youth mental health trajectories over time? RQ 2: Is there a reciprocal relationship between youth mental health problems and caregiver burden? RQ 2a: Do family processes mediate the association between caregiver burden and youth mental health problems? RQ 3: How do caregivers experience their children's return to home care? RQ 3a: What challenges and needs do caregivers report? RQ 3b: What types of follow-up services do families receive and/or have access to? RQ 3c: How do caregivers cope with ongoing difficulties in the post-discharge period?

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* primary caregiver of a child or adolescent aged 7-21 years of any gender who received inpatient treatment in a psychiatric institution in Germany, Austria, or Switzerland (min. 24 h stay) within the past month (regardless of the diagnosis or the reason for the treatment, respectively)
* lived with the child or adolescent in the same household since discharge

Exclusion Criteria:

* another caregiver of the same child has already participated in the study
* insufficient knowledge of German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary caregivers (parents or guardians regardless of the biological relationship to the child) of children and adolescents who received inpatient psychiatric treatment
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Inpatient readmission | Within 6 months
  Occurrence (and admission date) of inpatient mental health treatment after discharge
Youth mental health | Change from baseline (T0) to 3-month (T1) and 6-month (T2) follow-up
  Caregiver-reported youth internalizing and externalizing problems (assessed using the Pediatric Symptom Checklist)

SECONDARY OUTCOMES:
Youth health-related quality of life | Change from baseline (T0) to 3-month (T1) and 6-month (T2) follow-up
  Quality of life related to self-esteem, school, and peer relationships (assessed using the KINDL-R)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Zemp, Professor, Principal Investigator — University of Vienna